CLINICAL TRIAL: NCT07013864
Title: Staphylococcus Haemolyticus in the Neonatal Intensive Care Unit of CHSD in 2023: Analysis and Trends
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0086_NEONATOLOGIE
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Staphylococcus Haemolyticus; Staphylococcal Infections; Sepsis; Catheter-Related Infections; Infant, Newborn; Intensive Care Units, Neonatal; Cross Infection; Drug Resistance, Bacterial
MeSH Terms: conditions — Staphylococcal Infections; Sepsis; Catheter-Related Infections; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at cases of Staphylococcus haemolyticus infections in newborns hospitalized in the Neonatal Intensive Care Unit (NICU) at the Saint-Denis Hospital in 2023. Researchers reviewed the medical records of 28 infants who had this bacteria found in their blood or catheter cultures. The goal is to understand whether these infections have increased and how they affected the babies' health.

ELIGIBILITY:
Inclusion Criteria:

* Newborns in 2023
* hospitalized in the Neonatal and Neonatal Resuscitation department of the Saint-Denis
* At least one isolation of S. haemolyticus in blood cultures or catheter cultures

Exclusion Criteria:

- No exclusion criteria

Max Age: 2 Months | Sex: All
Age Groups: Child
Study Population: The inclusion criteria were all newborns in 2023, hospitalized in the Neonatal and Neonatal Resuscitation department of the Saint-Denis Hospital Centre with at least one isolation of S. haemolyticus in blood cultures or catheter cultures.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Staphylococcus haemolyticus Infections Associated with Central Venous Catheters (CVCs) | January 1, 2023 - December 31, 2023

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France